CLINICAL TRIAL: NCT07016464
Title: A Phase 1, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study of REM0045392 to Evaluate Pharmacokinetics, Pharmacodynamics, Safety, Tolerability, and Food Effect in Healthy Male Participants and in a Panel of Healthy Elderly Participants (Both Sexes)
Brief Title: A Study to Investigate Safety, Tolerability and Pharmacokinetics of REM0045392 Compared With Placebo in Healthy Participants.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: reMYND (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REMAD-04
Record Dates: First submitted 2025-05-23; First posted 2025-06-11 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Part 1 SAD - Panel A Treatment Period 1 (Experimental)
  Interventions: Drug: REM0045392; Drug: Placebo
- Part 1 SAD - Panel B Treatment Period 1 (Experimental)
  Interventions: Drug: REM0045392; Drug: Placebo
- Part 1 SAD - Panel A Treatment Period 2 (Experimental)
  Interventions: Drug: REM0045392; Drug: Placebo
- Part 1 SAD - Panel B Treatment Period 2 (Experimental)
  Interventions: Drug: REM0045392; Drug: Placebo
- Part 1 SAD - Panel A Treatment Period 3 (Experimental)
  Interventions: Drug: REM0045392; Drug: Placebo
- Part 1 SAD - Panel B Treatment Period 3 (Experimental)
  Interventions: Drug: REM0045392; Drug: Placebo
- Part 1 SAD - Panel A Treatment Period 4 (Experimental)
  Interventions: Drug: REM0045392; Drug: Placebo
- Part 1 SAD - Panel B Treatment Period 4 (Experimental)
  Interventions: Drug: REM0045392; Drug: Placebo
- Part 2 MAD - Panel C (Experimental)
  Interventions: Drug: REM0045392; Drug: Placebo
- Part 2 MAD - Panel D (Experimental)
  Interventions: Drug: REM0045392; Drug: Placebo
- Part 2 MAD - Panel E (Experimental)
  Interventions: Drug: REM0045392; Drug: Placebo
- Part 3 Elderly - Panel G (Experimental)
  Interventions: Drug: REM0045392; Drug: Placebo
- Part 2 MAD - Panel F (optional) (Experimental)
  Interventions: Drug: REM0045392; Drug: Placebo
- Part 3 Elderly - Panel H (optional) (Experimental)
  Interventions: Drug: REM0045392; Drug: Placebo

INTERVENTIONS:
Drug: REM0045392 — Liquid formulation
Drug: Placebo — Liquid formulation

SUMMARY:
This study is testing if the medicine REM0045392 is safe and well-tolerated. It also looks at whether food affects how the medicine works.

The medicine will be tested in Healthy men (Part 1 and 2) and Healthy Older men and women (Part 3).

Participants will take the medicine once (in Part 1) or during 14 days (in Part 2 and 3), with increasing doses.

REM0045392 is being developed as a treatment for Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male participants between 18 and 55 years of age, inclusive, at screening. For Part 3: male and females participants, aged between 65 and 85 years of age, inclusive, at screening
2. Otherwise healthy with no clinically significant abnormalities as determined by medical history, coagulation, blood chemistry assessments, hematologic assessments, and urinalysis at screening; and physical examination, measurement of vital signs and ECG at screening and Day 1 predose (of the first treatment period, if applicable).

   Note: Isolated out-of-range values judged by the investigator (or designated physician) to be of no clinical significance can be allowed. This determination must be recorded in the electronic source (eSource) system.

   For Part 3: elderly participants should be healthy for age. Mild and controlled comorbidities can be allowed at the discretion of the Investigator - as long as they do not interfere with the objectives of the study
3. Have a body weight in the range of 50 to 100 kg, inclusive, at screening. Have a body mass index (BMI) of 19.0 to 30.0 kg/m2, inclusive, at screening.

   For Part 3: have a BMI of 19.0 to 32.0 kg/m2, inclusive, at screening
4. Agree to abstain from alcohol intake 24 hours before administration of investigational product, during the in-patient period of the study, and 24 hours prior to all other out patient clinic visits.
5. Agree not to use prescription medications within 14 days prior to first investigational product administration and through the end of the study, unless approved by the investigator.

   For Part 3: elderly participants can be allowed to take their chronic medication (> 3 months stable dose) if this medication does not interfere with the absorption, distribution and elimination of the study drug.
6. Agree not to use over-the-counter medications (including corticosteroids, Aspirin, decongestants, antihistamines, and other non-steroidal anti-inflammatory drugs [NSAIDs]), and herbal medication (including herbal tea, St. John's Wort), within 14 days prior to the first investigational product administration through the end of the study, unless approved by the investigator.
7. Have signed the Informed Consent Form (ICF) voluntarily before any study related procedure is performed, indicating that the participant understands the purpose of, and procedures required for the study and is willing to participate in the study.
8. Male participants who are sexually active with a female partner must agree to the use of an effective method of birth control throughout the study and until 90 days after the last administration of investigational product. Sperm donation is also not allowed from the first administration until 90 days after the last administration of investigational product.

Note: Medically acceptable method of contraception that may be used by the participant includes vasectomy for male participants and for non-vasectomized male participants having a female partner of childbearing potential acceptable options includes using a condom in combination with one of the following: combined oral contraceptive, contraceptive injection, intrauterine device, levonorgestrel implant, or being surgically sterile. For male participants having a female pregnant partner, a condom must be used.

For Part 3: female participants should be postmenopausal as defined as spontaneous amenorrhea for more then 12 consecutive months; or spontaneous amenorrhea for less then 6 months with biochemical criteria of menopause (follicle-stimulating hormone >40 IU/L) or surgically sterile.

Exclusion Criteria:

1. Currently have or have a history of any clinically significant medical illness or medical disorders the investigator considers should exclude the participant, including (but not limited to) cardiovascular disease, neuromuscular disease, hematological disease, immune deficiency state, respiratory disease, hepatic or gastrointestinal disease, neurological or psychiatric disease, ophthalmological disorders, neoplastic disease, renal or urinary tract diseases, diseases affecting bone mineral density, endocrine disease, or dermatological disease.
2. Have a clinically significant or chronic infection or diagnosed latent infection.
3. Significant acute illness within 7 days prior to the first investigational product administration or have had a major illness or hospitalization within 1 month prior to the first investigational product administration.
4. For CSF collection:

   1. Lower back surgery in the past interfering with lumbar puncture
   2. History of severe Post Dural Puncture Headache requiring blood patch (PDPH)
   3. History or indications of elevated intracranial pressure as observed (fundoscopy)
5. Any of the following findings on resting ECG:

   1. QT interval corrected for heart rate (HR) using Fridericia's formula (QTcF) > 450 ms (males) or < 300 ms at screening or baseline visit (Day 1 pre dose).
   2. Notable resting bradycardia (HR < 40 bpm) or tachycardia (HR > 100 bpm) at screening or baseline visit (Day 1 pre-dose).
   3. Family history of congenital long QT syndrome or sudden death.
   4. Screening or baseline (Day 1 pre-dose) ECG with QRS and/or T wave judged to be unfavorable for a consistently accurate QT measurement (e.g., neuromuscular artifact that cannot be readily eliminated, arrhythmia, indistinct QRS onset, low amplitude T wave, merged T and U waves, prominent U waves).
   5. Evidence of atrial fibrillation, atrial flutter, complete left or right bundle branch block (LBBB/RBBB), incomplete LBBB, incomplete RBBB, Wolf Parkinson White syndrome, or cardiac pacemaker at screening or baseline visit (Day 1 pre-dose) (note: a first-degree heart block with PR not exceeding 250 ms can be allowed).

      For Part 3: in elderly participants:
   6. QTcF > 450 ms (males); > 470 ms (females) or < 300 ms at screening or baseline visit (Day 1 pre dose).
   7. Notable resting bradycardia (HR < 45 bpm) or tachycardia (HR > 100 bpm) at screening or baseline visit (Day 1 pre-dose).
   8. Family history of congenital long QT syndrome or sudden death.
   9. Wolff Parkinson White syndrome, complete LBBB (note: a first-degree heart block with PR not exceeding 250 ms, treated atrial fibrillation /flutter and incomplete LBBB can be allowed).
6. Have an estimated glomerular filtration rate (eGFR) using the Chronic Kidney Disease - Epidemiology Collaboration (CKD-EPI) method of < 80 mL/min/1.73 m².

   For Part 3: elderly participants have an eGFR (CKD-EPI) <60 mL/min/1.73 m². In case of an abnormal result, recheck is authorized if needed and this recheck can consist of a 24h urine collection to measure real creatinine clearance when deemed necessary.
7. Systolic blood pressure (SBP) greater than 140 or less than 90 mmHg, and diastolic blood pressure (DBP) greater than 90 or less than 45 mm Hg For Part 3: in elderly participants: SBP greater than 160 or less than 90 mmHg, and DBP greater than 95 or less than 45 mm Hg
8. Major or traumatic surgery within 12 weeks of screening.
9. Any participant who plans to undergo elective surgery within 4 weeks prior to the first investigational product administration and through the end of the study.
10. Positive serology test for human immunodeficiency virus (HIV) type 1 and 2 antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibodies at screening.
11. Recent history (within the previous 6 months from screening) of alcohol or drug abuse.
12. Active smoker and/or has used nicotine or nicotine-containing products (including e-cigarettes or the equivalent of e-cigarettes) within the past 6 months before the first investigational product administration.
13. Have positive urine toxicology screen at screening or Day -1 for substances of abuse including amphetamines, benzodiazepine, cocaine, opiates, methadone, cannabinoids, and tricyclic antidepressants.

    Note: Participants should not consume poppy seeds within 24 hours before screening and before each urine drug screening because this can falsify the results of the opiate urine drug test.
14. Have a positive alcohol breath test at screening or Day -1.
15. Consumes, on average, more than approximately 500 mg/day of caffeine (as contained in 5 cups of tea or coffee or 8 cans of soda or other caffeinated products per day) at screening.
16. Donated blood within 90 days prior to first investigational administration.
17. Have a history of active drug and/or food allergy or other active allergic disease requiring the constant use of medications, or a history of severe allergic reaction, angioedema or anaphylaxis at screening.
18. Received any other experimental therapy or new investigational agent within 30 days or 5 half-lives (whichever is longer) of the first investigational product administration.
19. Treatment with any medication (including over-the-counter and/or prescription medication, dietary supplements, nutraceuticals, vitamins and/or herbal supplements) except occasional paracetamol (maximum dose of 2 g/day and maximum of 10 g/2 weeks), in the last 2 weeks or 5 half-lives of the drug, whichever is longer, prior to the first dosing of investigational product For Part 3: elderly participants taking the following prohibited medications/substances: Strong Cytochrome (CYP) 3A4-1A2-2D6 inhibitors (Wash out prior to Baseline 30 days or 5 half-lives, whichever is longer), and sensitive CYP2B6 -2D6 substrates (assessed on a case-by-case basis)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Related Adverse Events | Throughout the study, until 7-10 days post last dose
  To assess the safety and tolerability of REM0045392

SECONDARY OUTCOMES:
Assessment of pharmacokinetics (PK) in blood following single and multiple ascending oral dose administration | Up to 48 hours after last intervention
  Area under curve (AUC) in plasma
Assessment of pharmacokinetics (PK) in blood following single and multiple ascending oral dose administration | Up to 48 hours after last intervention
  Maximum concentration (Cmax) in plasma
Assessment of pharmacokinetics (PK) in blood following single and multiple ascending oral dose administration | Up to 48 hours after last intervention
  Time to peak drug concentration (Tmax) in plasma
Assessment of pharmacokinetics (PK) in blood following single and multiple ascending oral dose administration | Up to 48 hours after last intervention
  Half-life in plasma
Assessment of pharmacokinetics (PK) in blood following single and multiple ascending oral dose administration | Up to 48 hours after last intervention
  Clearance (CL/F) in plasma
Assessment of pharmacokinetics (PK) in blood following single and multiple ascending oral dose administration | Up to 48 hours after last intervention
  Volume of distribution (V/F) in plasma
Assessment of pharmacokinetics (PK) in blood following single and multiple ascending oral dose administration | Up to 48 hours after last intervention
  Peak to trough fluctuation ratio in plasma
Assessment of pharmacokinetics (PK) in blood following single and multiple ascending oral dose administration | Up to 48 hours after last intervention
  Accumulation index in plasma
Concentrations of REM0045392 measured in CSF samples | Up to 24h after study intervention
Assessment of the effect of REM0045392 on the QT interval on ECG | Up to 48h after last intervention
  QTc changes in function of observed plasma concentrations of REM0045932

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Belgium NV - Clinical Pharmacology Unit, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No